CLINICAL TRIAL: NCT05649293
Title: Assesment of Vitamin B6 Level in Patients With Major Depressive Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omnia Abd El Nasser Badry, doctor, Assiut University
Other Study IDs: vitamin b6 & depression
Record Dates: First submitted 2022-12-05; First posted 2022-12-14 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Vitamin b6 Level & Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- major depressive disorder patients: patient diagnosed with major depression for first time
  Interventions: Other: measure vitamin b6 in serum
- depression free persons: healthy persons
  Interventions: Other: measure vitamin b6 in serum

INTERVENTIONS:
Other: measure vitamin b6 in serum — * Vitamin B6 levels can be determined by using Enzyme- linked Immuno-sorbent Assay Kit For vitamin B6 . or Chemiluminescence Immunoassays (CLIA) .
  * Venous blood samples will be taken from each patient. Use a serum separator tube and allow samples to clot for 10-20 minutes at room temperature and then centrifuged for 20 minutes at speed of 2000-3000 rpm (round per minute).
  * Remove supernatant, if precipitation appeared, Centrifuge again.
  * Extract as soon as possible after Samples collection, and should be tested as soon as possible after the extraction.
  * If not, samples must be stored in aliquot at -20°C (≤ 1 month) or -80°C (≤ 2 months) to avoid loss of bioactivity and contamination.
  * Hemolyzed Sample will be avoided , as hemolysis will interfere with the results .

SUMMARY:
Estimation of vitamin B 6 levels in diagnosed major depressive disorder patients and their relation to the severity of the disease

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a chronic health condition with significant consequences for health care costs, disability, quality of life, medical morbidity, and mortality. The World Health Organization (WHO) has considered depression as the leading cause of disability, a major contributor to overall global burden of disease . The core symptoms of depression are low mood and loss of interest or enjoyment in usually pleasurable activities. Associated symptoms include disturbances to sleep and appetite, reduced energy and concentration, negative thoughts of guilt or worthlessness and suicidal ideation. The International Statistical Classification of Diseases & Related Health Problems (ICD-10) states that for a diagnosis of depression at least five symptoms need to be present, including at least one of the core symptoms, at an intensity that causes functional impairment and for a minimum duration of 2 weeks.

Vitamin B6 (Pyridoxine) is a water-soluble compound that comprises three different pyridine derivatives, pyridoxine, pyridoxal, and pyridoxamine, of which PLP(pyridoxal phosphate) is the biologically most active form. The coenzyme PLP is an essential cofactor for amino acid decarboxylases involved in the synthesis of neurotransmitters implicated in depression, including dopamine, norepinephrine ,serotonin or 5-hydroxytryptamine (5-HT), and γ-amino butyric acid (GABA). it prevents the accumulation of neurotoxic intermediates produced during tryptophan metabolism, acting as a cofactor in the metabolism of tryptophan through the kynurenine aminotransferase and kynureninase enzymes. Inadequate intake of vitamin B6 has recently been linked to an increased risk of anxiety and depression in a cross-sectional study of over 3,000 individuals.

ELIGIBILITY:
Inclusion Criteria:

* All participants must fulfill the following inclusion criteria;

  1. Patients diagnosed newly as major depressive disorder according to DSM-5( Diagnostic and Statistical Manual ) and (APA 2013) .
  2. Aged at least 18 years of both sex .
  3. Able to give informed consent .

Exclusion Criteria:

1. Patients have Comorbidity with other psychiatric disorders .
2. Patients have chronic medical conditions , chronic debilitating or nutritional disorders .
3. for control , Patients with any psychiatric disorders .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 94 participants divided into 47 patients diagnosed with major depressive disorder and 47 of normal population as control.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assesment of vitamin B6 level in patients with Major Depressive Disorder | baseline
  Estimation of vitamin B 6 levels in diagnosed major depressive disorder patients and their relation to the severity of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdel Rahman, Prof, Study Director — Assiut University; Romany H Gabra, dr, Study Director — Assiut University

REFERENCES:
- [Background] Hvas AM, Juul S, Bech P, Nexo E. Vitamin B6 level is associated with symptoms of depression. Psychother Psychosom. 2004 Nov-Dec;73(6):340-3. doi: 10.1159/000080386. PMID 15479988
- [Background] Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). J Clin Psychiatry. 2015 Feb;76(2):155-62. doi: 10.4088/JCP.14m09298. PMID 25742202
- [Background] Coppen A, Bailey J. Enhancement of the antidepressant action of fluoxetine by folic acid: a randomised, placebo controlled trial. J Affect Disord. 2000 Nov;60(2):121-30. doi: 10.1016/s0165-0327(00)00153-1. PMID 10967371
- [Background] Eisenberg DM, Davis RB, Ettner SL, Appel S, Wilkey S, Van Rompay M, Kessler RC. Trends in alternative medicine use in the United States, 1990-1997: results of a follow-up national survey. JAMA. 1998 Nov 11;280(18):1569-75. doi: 10.1001/jama.280.18.1569. PMID 9820257
- [Background] Arevalo SP, Scott TM, Falcon LM, Tucker KL. Vitamin B-6 and depressive symptomatology, over time, in older Latino adults. Nutr Neurosci. 2019 Sep;22(9):625-636. doi: 10.1080/1028415X.2017.1422904. Epub 2018 Jan 16. PMID 29338677
- [Background] Moore K, Hughes CF, Hoey L, Ward M, Cunningham C, Molloy AM, Strain JJ, McCarroll K, Casey MC, Tracey F, Laird E, O'Kane M, McNulty H. B-vitamins in Relation to Depression in Older Adults Over 60 Years of Age: The Trinity Ulster Department of Agriculture (TUDA) Cohort Study. J Am Med Dir Assoc. 2019 May;20(5):551-557.e1. doi: 10.1016/j.jamda.2018.11.031. Epub 2019 Jan 25. PMID 30692033